CLINICAL TRIAL: NCT05890001
Title: A Study to Evaluate the Long-Term Safety of BLI5100 in Patients With Gastroesophageal Reflux Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BLI5100-303
Record Dates: First submitted 2023-05-05; First posted 2023-06-05 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Non-erosive Reflux Disease; Erosive Esophagitis
MeSH Terms: conditions — Non-Erosive Reflux Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BLI5100 Low Dose (Experimental): Patients will take BLI5100 Low Dose once daily, orally, for up to 29 weeks.
  Interventions: Drug: BLI5100
- BLI5100 High Dose (Experimental): Patients will take BLI5100 High Dose once daily, orally, for up to 29 weeks.
  Interventions: Drug: BLI5100

INTERVENTIONS:
Drug: BLI5100 — Patients will take BLI5100 once daily, orally, for up to 29 weeks.

SUMMARY:
The objective of this study is to evaluate the safety of up to 12 months (52 weeks) of once daily oral administration of BLI5100 in patients with non-erosive reflux disease (NERD) or healed erosive esophagitis (EE).

ELIGIBILITY:
Inclusion Criteria:

1. Have completed the BLI5100-301 or BLI5100-302 study with no serious AE (SAE) related to study drug and no major Protocol Deviations;
2. Able to understand and comply with the protocol requirements;
3. Willing and able to provide written informed consent at Screening;
4. Is a female of non-childbearing potential, or If a female of childbearing potential, agrees to use an acceptable form of birth control and avoid egg donation from the Screening Visit until 6 months after the last dose of study drug;
5. If a male, agrees to use an acceptable form of birth control from the Screening Visit until 3 months after the last dose of study drug;
6. If a male, agrees to abstain from sperm donation through 3 months after administration of the last dose of study drug;
7. Have documented healed EE (BLI5100-301 study patients only).

Exclusion Criteria:

1. History of alcoholism, or substance abuse/addiction in the year before enrollment in the BLI5100-301 and BLI5100-302 studies;

   * Note: Patients on prescribed opioids are eligible to participate if they have been on a stable dose for the duration of the BLI5100-301 and BLI5100-302 studies.
   * Note: Retesting of a positive urine drug screen requires Medical Monitor approval. Positive urine drug screen for all drugs will require verification of prescription for the positive tested substance.
2. A diagnosis of manic-depression, anxiety disorder, panic disorder, somatoform disorder, personality disorder, or other psychological disorder is exclusionary, unless the patient is asymptomatic and well-controlled. Stable treatment, including non-medical therapy, is preferred, but minor adjustments can be made and should be consulted with the Medical Monitor;
3. Current use of antipsychotics, antidepressants, anxiolytics, or prescription sleeping medications, with the exception of a stable dose for the duration of the BLI5100-301 and BLI5100-302 studies;
4. Requirement of persistent (>3 times per week for >30 days) use of non-steroidal anti-inflammatory drugs (NSAIDs) during the course of the study;

   o Note: Low-dose (≤100 mg/day) aspirin is allowed provided that it has been used for prophylaxis prior to study participation.
5. If a female, is pregnant, breastfeeding, or planning to become pregnant during the study or within 6 months after the last dose of study drug;
6. Abnormal laboratory results with clinical relevance at Screening as follows:

   * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), or alkaline phosphatase level of ≥2 × upper limit of normal (ULN);
   * Total bilirubin level of ≥2 × ULN, unless Gilbert's syndrome is confirmed when direct bilirubin is ≤0.3 mg/dL;
   * Estimated glomerular filtration rate <30 mL/min.
   * Note: A lab value obtained during the Screening period may be retested once with Medical Monitor approval.
7. Abnormal ECG of clinical significance;
8. Involvement in another clinical study (other than BLI5100-301 and BLI5100-302 studies) within 4 weeks of initiation of study drug;
9. Any other clinically relevant condition that would confound study endpoints or adversely affect patient compliance with the study procedures in the medical judgment of the Investigator or Medical Monitor based on previous medical history or findings on Screening assessments.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
Frequency of treatment-emergent adverse events | 31 Weeks

CONTACTS AND LOCATIONS:
Locations (60):
- United States (60):
  - Research Site 24, Huntsville, Alabama
  - Research Site 62, Phoenix, Arizona
  - Research Site 27, Tucson, Arizona
  - Research Site 87, Little Rock, Arkansas
  - Research Site 117, North Little Rock, Arkansas
  - Research Site 94, Chula Vista, California
  - Research Site 10, Huntington Park, California
  - Research Site 55, La Mesa, California
  - Research Site 72, Los Angeles, California
  - Research Site 54, Los Angeles, California
  - Research Site 13, Santa Ana, California
  - Research Site 41, Santa Maria, California
  - Research Site 108, Cooper City, Florida
  - Research Site 91, Doral, Florida
  - Research Site 78, Homestead, Florida
  - Research Site 23, Maitland, Florida
  - Research Site 38, Miami, Florida
  - Research Site 43, Miami, Florida
  - Research Site 67, Miami, Florida
  - Research Site 92, Miami, Florida
  - Research Site 71, Miami, Florida
  - Research Site 42, Miami Lakes, Florida
  - Research Site 17, New Port Richey, Florida
  - Research Site 90, Ocoee, Florida
  - Research Site 05, Palmetto Bay, Florida
  - Research Site 11, Sunrise, Florida
  - Research Site 46, Viera, Florida
  - Research Site 59, Sandy Springs, Georgia
  - Research Site 01, Gurnee, Illinois
  - Research Site 02, Oak Lawn, Illinois
  - Research Site 45, Houma, Louisiana
  - Research Site 12, Marrero, Louisiana
  - Research Site 48, Metairie, Louisiana
  - Research Site 34, New Orleans, Louisiana
  - Research Site 111, Chesterfield, Missouri
  - Research Site 06, Las Vegas, Nevada
  - Research Site 64, Reno, Nevada
  - Research Site 35, Brooklyn, New York
  - Research Site 07, Great Neck, New York
  - Research Site 28, Hartsdale, New York
  - Research Site 49, New York, New York
  - Research Site 40, Rochester, New York
  - Research Site 75, Fayetteville, North Carolina
  - Research Site 20, Columbus, Ohio
  - Research Site 88, Columbus, Ohio
  - Research Site 109, Mentor, Ohio
  - Research Site 110, Westlake, Ohio
  - Research Site 60, Nashville, Tennessee
  - Research Site 103, Nashville, Tennessee
  - Research Site 100, Bellaire, Texas
  - Research Site 98, Dallas, Texas
  - Research Site 99, Forney, Texas
  - Research Site 29, Lewisville, Texas
  - Research Site 32, Pearland, Texas
  - Research Site 30, Red Oak, Texas
  - Research Site 22, San Antonio, Texas
  - Research Site 26, San Antonio, Texas
  - Research Site 21, San Antonio, Texas
  - Research Site 65, Sandy City, Utah
  - Research Site 16, South Ogden, Utah

IPD SHARING:
Plan to Share IPD: No